CLINICAL TRIAL: NCT00153894
Title: Pilot Study of the Effects of an Exercise Intervention on Insulin Levels in Breast Cancer Survivors
Brief Title: Effects of Exercise Intervention on Insulin Levels in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-327
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer survivor; Insulin levels; exercise regimen; endurance training; strength training
MeSH Terms: conditions — Breast Neoplasms | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Immediate Exercise
  Interventions: Behavioral: Strength training; Behavioral: Endurance training
- Group B (Active Comparator): Delayed Exercise (delay by 16 weeks)
  Interventions: Behavioral: Strength training; Behavioral: Endurance training

INTERVENTIONS:
Behavioral: Strength training — One-on-One training with a personal trainer for 50 minutes twice a week using Nautilus machines for 16 weeks.
Behavioral: Endurance training — Cardiovascular training at home for 30 minutes three times per week for 16 weeks.

SUMMARY:
The purpose of this study is to determine whether an exercise program comprised of strength and endurance training will lower fasting insulin levels in a group of breast cancer survivors. Insulin may be involved in the risk of breast cancer recurrence.

DETAILED DESCRIPTION:
* All women taking part in this study will take part in an exercise program. Group A will start exercising immediately and Group B wil have a delay period of 16 weeks before starting to exercise so investigators can look at the changes in insulin levels that occur in a women who is not exercising.
* The exercise program will be made up of two parts: strength (or weight) training and cardiovascular exercise. The strength exercise will take place at a gym close to Dana-Farber Cancer Institute. Patients will work one on one with a personal trainer twice a week for 50 minutes. During each of these sessions, participants will have a brief warm up period and then will perform a series of Nautilus machine-based exercises under the guidance of the personal trainer. The goal of each session will be to increase strength by increasing weight lifted and repetitions.
* Participants will also do cardiovascular exercises on their own at home. Each participant will receive a pedometer and heart rate monitor. Women will be advised to exercise for at least 30 minutes three times per week on their own and will keep a journal recording how long and how intensively they exercised. Participants will receive weekly phone calls from the project manager to review the cardiovascular exercise.
* Women will undergo a series of measurements before and after the 16 week exercise intervention. They will be asked to fast for 12 hours prior to each of these measurement sessions. Measurements will include blood testing for insulin and glucose levels. Women will also be weighed, height will be measured, body composition will be computed using a noninvasive bioelectric impedance monitor, and hip/waist measurements will be taken. Group A participants will undergo testing at the time of enrolling in the study and after 16 weeks of exercise. Group B participants will undergo these tests after enrollment, after the 16 week waiting period and at the end of the exercise program.
* Participants will also complete two surveys by mail, 3 months and 9 months after completing the exercise portion of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of pathologically confirmed stage I-IIIa invasive breast cancer
* Adjuvant chemotherapy and/or radiation must be completed at least 3 months prior to enrollment
* Body mass index > 25 and/or a body composition analysis of >30

Exclusion Criteria:

* Patients taking herceptin
* Evidence of residual or distant disease
* Use of any medication expected to affect insulin levels
* Baseline exercise of more than 20 minutes two times per week
* Active malignancy
* Diabetes mellitus
* Heart disease or uncontrolled hypertension
* Presence of any condition that might be expected to impact a participant's ability to perform physical activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-12; Primary Completion 2006-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine whether strength and endurance training will lower fasting insulin levels in a group of breast cancer survivors. | 3 years

SECONDARY OUTCOMES:
To assess the compliance of a group of breast cancer survivors to a 16 week exercise intervention | 3 years
to determine whether a combination strength and endurance training intervention can increase strength and endurance by 25% over a 16 week training period | 3 years
to evaluate the impact of an exercise intervention on weight, waist-hip ratio and body composition in breast cancer survivors. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ligibel JA, Giobbie-Hurder A, Olenczuk D, Campbell N, Salinardi T, Winer EP, Mantzoros CS. Impact of a mixed strength and endurance exercise intervention on levels of adiponectin, high molecular weight adiponectin and leptin in breast cancer survivors. Cancer Causes Control. 2009 Oct;20(8):1523-8. doi: 10.1007/s10552-009-9358-3. Epub 2009 May 13. PMID 19434504
- [Result] Ligibel JA, Campbell N, Partridge A, Chen WY, Salinardi T, Chen H, Adloff K, Keshaviah A, Winer EP. Impact of a mixed strength and endurance exercise intervention on insulin levels in breast cancer survivors. J Clin Oncol. 2008 Feb 20;26(6):907-12. doi: 10.1200/JCO.2007.12.7357. PMID 18281663